CLINICAL TRIAL: NCT01541800
Title: A Feasibility Study of Circulating microRNAs as Disease Markers in Pediatric Cancers
Brief Title: Circulating microRNAs as Disease Markers in Pediatric Cancers
Status: Completed | Type: Observational
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 2010-14205
Record Dates: First submitted 2012-02-24; First posted 2012-03-01 (Estimated); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Leukemia; Lymphoma; Central Nervous System
MeSH Terms: conditions — Leukemia; Lymphoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood and cerebral spinal fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients: All children who are in treatment for leukemia, lymphoblastic lymphoma and central nervous system tumors between 3 years and 21 years of age

SUMMARY:
MicroRNAs are small molecules which have recently been discovered in cells. They are known to be responsible for the normal development of cells and when they are disrupted can contribute to the development of cancer. Many previous studies have been done evaluating the expression of microRNAs in normal tissues as well as a wide variety of cancers.

Recently, microRNAs from tumor cells have been detected circulating in the blood of patients with cancer. This presents a novel opportunity to use microRNAs in the blood as an early predictor of cancer as well as a marker of response to therapy. No previous studies have been performed evaluating microRNAs in the blood or cerebrospinal fluid of patients with childhood cancers. We propose a feasibility study to evaluate the presence of microRNAs in the blood and cerebrospinal fluid of patients with central nervous system tumors, leukemia and lymphoma who are currently on chemotherapy and undergoing blood draws, lumbar punctures and/or reservoir taps for routine clinical care. If we're able to identify circulating microRNAs in this population of pediatric patients, we will build upon this data in proposing a future study.

ELIGIBILITY:
Inclusion Criteria:

* All children who are in treatment for leukemia, lymphoblastic lymphoma and central nervous system tumors
* age: greater than 3 years and less than or equal to 21 years of age
* Patients must be in a phase of their treatment during which routine blood draws, lumbar punctures or CSF sampling from Ommaya reservoirs are required for treatment of their cancers.

Exclusion Criteria:

* Patients who have completed treatment and do not require routine blood draws and/or lumbar punctures
* Patients who are considered too ill to participate as determined by their treating physician
* Patients with a known genetic condition that predisposed them to the development of cancer.

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children who are in treatment for leukemia, lymphoblastic lymphoma and central nervous system tumors
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Determine if miRNAs are present in the blood of patients with pediatric cancers | 1 year
Determine if miRNAs are detectable in the CSF of patients with pediatric cancers. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Rishi Lulla, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Fernandez-L A, Northcott PA, Taylor MD, Kenney AM. Normal and oncogenic roles for microRNAs in the developing brain. Cell Cycle. 2009 Dec 15;8(24):4049-54. doi: 10.4161/cc.8.24.10243. Epub 2009 Dec 5. PMID 19901543
- [Background] Roth C, Rack B, Muller V, Janni W, Pantel K, Schwarzenbach H. Circulating microRNAs as blood-based markers for patients with primary and metastatic breast cancer. Breast Cancer Res. 2010;12(6):R90. doi: 10.1186/bcr2766. Epub 2010 Nov 3. PMID 21047409
- [Background] Taylor DD, Gercel-Taylor C. MicroRNA signatures of tumor-derived exosomes as diagnostic biomarkers of ovarian cancer. Gynecol Oncol. 2008 Jul;110(1):13-21. doi: 10.1016/j.ygyno.2008.04.033. PMID 18589210
- [Background] Lawrie CH, Gal S, Dunlop HM, Pushkaran B, Liggins AP, Pulford K, Banham AH, Pezzella F, Boultwood J, Wainscoat JS, Hatton CS, Harris AL. Detection of elevated levels of tumour-associated microRNAs in serum of patients with diffuse large B-cell lymphoma. Br J Haematol. 2008 May;141(5):672-5. doi: 10.1111/j.1365-2141.2008.07077.x. Epub 2008 Mar 3. PMID 18318758
- [Background] Huang Z, Huang D, Ni S, Peng Z, Sheng W, Du X. Plasma microRNAs are promising novel biomarkers for early detection of colorectal cancer. Int J Cancer. 2010 Jul 1;127(1):118-26. doi: 10.1002/ijc.25007. PMID 19876917
- [Background] Ng EK, Chong WW, Jin H, Lam EK, Shin VY, Yu J, Poon TC, Ng SS, Sung JJ. Differential expression of microRNAs in plasma of patients with colorectal cancer: a potential marker for colorectal cancer screening. Gut. 2009 Oct;58(10):1375-81. doi: 10.1136/gut.2008.167817. Epub 2009 Feb 6. PMID 19201770
- [Background] Heneghan HM, Miller N, Lowery AJ, Sweeney KJ, Kerin MJ. MicroRNAs as Novel Biomarkers for Breast Cancer. J Oncol. 2009;2009:950201. doi: 10.1155/2010/950201. Epub 2009 Jul 20. PMID 19639033
- [Background] Zhu W, Qin W, Atasoy U, Sauter ER. Circulating microRNAs in breast cancer and healthy subjects. BMC Res Notes. 2009 May 19;2:89. doi: 10.1186/1756-0500-2-89. PMID 19454029
- [Background] Wang K, Zhang S, Marzolf B, Troisch P, Brightman A, Hu Z, Hood LE, Galas DJ. Circulating microRNAs, potential biomarkers for drug-induced liver injury. Proc Natl Acad Sci U S A. 2009 Mar 17;106(11):4402-7. doi: 10.1073/pnas.0813371106. Epub 2009 Feb 25. PMID 19246379
- [Background] Ji X, Takahashi R, Hiura Y, Hirokawa G, Fukushima Y, Iwai N. Plasma miR-208 as a biomarker of myocardial injury. Clin Chem. 2009 Nov;55(11):1944-9. doi: 10.1373/clinchem.2009.125310. Epub 2009 Aug 20. PMID 19696117
- [Background] Ai J, Zhang R, Li Y, Pu J, Lu Y, Jiao J, Li K, Yu B, Li Z, Wang R, Wang L, Li Q, Wang N, Shan H, Li Z, Yang B. Circulating microRNA-1 as a potential novel biomarker for acute myocardial infarction. Biochem Biophys Res Commun. 2010 Jan 1;391(1):73-7. doi: 10.1016/j.bbrc.2009.11.005. Epub 2009 Nov 5. PMID 19896465
- [Background] Zhang H, Luo XQ, Zhang P, Huang LB, Zheng YS, Wu J, Zhou H, Qu LH, Xu L, Chen YQ. MicroRNA patterns associated with clinical prognostic parameters and CNS relapse prediction in pediatric acute leukemia. PLoS One. 2009 Nov 13;4(11):e7826. doi: 10.1371/journal.pone.0007826. PMID 19915715